CLINICAL TRIAL: NCT04617223
Title: Results of Endoscopic Sinus Surgery in Management of Ophthalmological Complications of Chronic Rhino Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Tadros, MD, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34062/8/20
Record Dates: First submitted 2020-10-13; First posted 2020-11-05 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other)
  Interventions: Procedure: Endoscopic sinus evacuation

INTERVENTIONS:
Procedure: Endoscopic sinus evacuation — Evacuation of the sinus by using endoscope

SUMMARY:
Investigate the clinical features of orbital complications of sinusitis in the Egyptian population, and observed that certain ophthalmological manifestations and outcomes were significantly associated with disease stage

DETAILED DESCRIPTION:
Retrospectively review of the medical records of all patients with orbital complications of paranasal sinusitis hospitalized at the ORL-HNS department at the University of Tanta between 2010 and 2020. Sex, age, symptoms, history, ophthalmological findings, laboratory and imaging findings, treatments, and outcomes were analyzed by staging.

The data that will be retrieved from the medical records including:

1. History taking including personal present and previous medical history.
2. General examination
3. Oto-rhinolaryngological clinical examination
4. Routine preoperative laboratory investigations (e.g. complete total and differential blood count, blood sugar, coagulation profile, and renal and liver function)
5. Diagnostic nasal Endoscopy with zero and/or a 30-degree telescope.
6. CT paranasal sinuses with contrast, fine cuts in coronal axial, and sagittal planes.
7. The type of intervention whether medical or surgical. 8- Culture results, treatments, hospital stay durations, and outcomes.

Ophthalmology data collection:

1. Visual acuity (onset of decrease) (unilateral or bilateral) ant its improvement after sinus surgery
2. Presence or absence of double vision (Diplopia)
3. Ocular motility and if its associated with pain
4. Proptosis (present or absent) and calculate the degree and direction
5. Ptosis (present or absent)
6. Pupil reactivity
7. Fundus examination to exclude optic nerve neuropathy
8. Association between ocular pain and headache and its improvement after surgery
9. CT data collection (CT orbit, MRI of sinus and head)
10. Fundus photography after surgery to see improvement of optic nerve neuropathy if present

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with preseptal/orbital inflammation secondary to acute (<1 month), subacute (1±3 months), or chronic sinusitis (>3 months) of bacterial, fungal or unidentified pathogens

Exclusion Criteria:

* Patients with chronic rhinosinusitis without orbital complication, Systemic diseases that affect the paranasal sinuses and the orbit e.g autoimmune diseases, lymphoma, leukaemia, Sinus or orbital malignancy, Data is missed from the charts

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
observe improvement of ophthalmological manifestation after surgical intervention | 1 month
  Measure the visual acuity by using Snellen chart and LogMAR chart (Logarithm of the minimum angle of resolution ) chart
  The Minimum number of snellen chart is 6/60 and maximum number is 6/6, The Minimum number of LogMAR chart is 1.0 and maximum number is - 0.1, The higher number means better vision
Improvement of the degree of proptosis after surgery | 1 month
  Decrease the degree of proptosis in millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Garbeia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 month
Access Criteria: link

REFERENCES:
- [Result] Hastan D, Fokkens WJ, Bachert C, Newson RB, Bislimovska J, Bockelbrink A, Bousquet PJ, Brozek G, Bruno A, Dahlen SE, Forsberg B, Gunnbjornsdottir M, Kasper L, Kramer U, Kowalski ML, Lange B, Lundback B, Salagean E, Todo-Bom A, Tomassen P, Toskala E, van Drunen CM, Bousquet J, Zuberbier T, Jarvis D, Burney P. Chronic rhinosinusitis in Europe--an underestimated disease. A GA(2)LEN study. Allergy. 2011 Sep;66(9):1216-23. doi: 10.1111/j.1398-9995.2011.02646.x. Epub 2011 May 24. PMID 21605125
- [Result] Shi JB, Fu QL, Zhang H, Cheng L, Wang YJ, Zhu DD, Lv W, Liu SX, Li PZ, Ou CQ, Xu G. Epidemiology of chronic rhinosinusitis: results from a cross-sectional survey in seven Chinese cities. Allergy. 2015 May;70(5):533-9. doi: 10.1111/all.12577. Epub 2015 Mar 4. PMID 25631304
- [Result] Chang YS, Chen PL, Hung JH, Chen HY, Lai CC, Ou CY, Chang CM, Wang CK, Cheng HC, Tseng SH. Orbital complications of paranasal sinusitis in Taiwan, 1988 through 2015: Acute ophthalmological manifestations, diagnosis, and management. PLoS One. 2017 Oct 3;12(10):e0184477. doi: 10.1371/journal.pone.0184477. eCollection 2017. PMID 28972988